CLINICAL TRIAL: NCT04457648
Title: Randomized Assessor Masked Trial Comparing Manuka Honey Eye Drops to Conventional Treatment of Meibomian Gland Dysfunction Related Dry Eye Disease.
Brief Title: Manuka Honey Eye Drops VS Conventional Treatment of Meibomian Gland Dysfunction Related Dry Eye Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Anita Li, Principal Investigator, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MGD1
Record Dates: First submitted 2020-06-26; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Meibomian Gland Dysfunction
MeSH Terms: conditions — Meibomian Gland Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional (Placebo Comparator)
  Interventions: Device: systane eye drops
- Manuka Honey (Active Comparator)
  Interventions: Device: manuka honey 16% eye drops ( Optimel )

INTERVENTIONS:
Device: manuka honey 16% eye drops ( Optimel ) — 16% manuka honey eye drops, australian FDA approved
  Arms: Manuka Honey
Device: systane eye drops — systane lubricant eye drops
  Arms: Conventional

SUMMARY:
Assessor-masked (Single blind, randomized controlled trial comparing the conventional treatment group to an interventional group using 16% Manuka Honey topical eye drops.

DETAILED DESCRIPTION:
Purpose To evaluate the effects of conventional treatment compared to use of Manuka Honey eye drops in the treatment of meibomian gland dysfunction related dry eye disease.

Design Assessor-masked (Single blind, randomized controlled trial comparing the conventional treatment group to an interventional group using 16% Manuka Honey topical eye drops.

Methods Patients were randomized into two groups, one group given conventional treatment for meibomian gland dysfunction. The other group was given additional manuka honey 16% eye drops which are registered as a medical device by the australian FDA. SPEED score was taken at baseline and upon follow up. Multiple parameters were graded from slit lamp examination by a masked assessor. Results were compared from baseline to follow up date 3 weeks later.

ELIGIBILITY:
Inclusion Criteria:

* meibomian gland dysfunction stage 2-4

Exclusion Criteria:

* <18 years old Unable to consent Recent ophthalmic surgery <6m Abnormalities of lid position Allergy to honey/bee products Contact lens wearers Patients on long term topical medications apart from lubricants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
speed score | 3 weeks
  questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- chinese university of Hong kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Yes
protocol
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 6 months after completion for 6 months

REFERENCES:
- [Derived] Li AL, Li SL, Kam KW, Young AL. Randomised assessor-masked trial evaluating topical manuka honey (Optimel) in treatment of meibomian gland dysfunction. Br J Ophthalmol. 2022 Jun;106(6):777-780. doi: 10.1136/bjophthalmol-2020-317506. Epub 2021 Jan 8. PMID 33419788